CLINICAL TRIAL: NCT06448845
Title: A Comparative Study Between Arm Intravenous Regional Anesthesia Versus Forearm Intravenous Regional Anesthesia in Patients Undergoing Hand and Wrist Surgery. A Randomized Comparative Prospective Clinical Study
Brief Title: A Comparative Study Between Arm Intravenous Regional Anesthesia Versus Forearm Intravenous Regional Anesthesia in Patients Undergoing Hand and Wrist Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD 148/2023
Record Dates: First submitted 2024-05-12; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Intravenous Anesthetic Agent Overdose; Hand Injury Wrist
Keywords: Forearm Tourniquet, Intravenous Regional Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Arm IVRA) 70 patients (Active Comparator): After placement of the upper arm and forearm tourniquets and exsanguination of the limb distal to the cuff by applying an Esmarch's bandage starting from the fingertips, the arm tourniquet cuff is inflated to a pressure of 250 mmHg. The double arm cuff pneumatic pressure tourniquet is placed immediately above the elbow crease and on the top of a circumferentially placed cotton cast padding before inflation.
  Interventions: Procedure: Arm intravenous regional anesthesia
- Group F (Forearm IVRA) 70 patients (Active Comparator): After placement of the forearm double tourniquet and exsanguination of the limb distal to the cuff by applying an Esmarch's bandage starting from the fingertips, the forearm tourniquet cuff is inflated to a pressure of 250 mmHg. The forearm tourniquet will be placed 5 cm distal to the medial epicondyle of the humerus and on the top of a circumferentially placed cotton cast.
  Interventions: Procedure: Forearm IVRA block

INTERVENTIONS:
Procedure: Arm intravenous regional anesthesia — After placement of the upper arm and forearm tourniquets and exsanguination of the limb distal to the cuff by applying an Esmarch's bandage starting from the fingertips, the arm tourniquet cuff is inflated to a pressure of 250 mmHg. The double arm cuff pneumatic pressure tourniquet is placed immediately above the elbow crease and on the top of a circumferentially placed cotton cast padding before inflation. Subsequently, tourniquet failure is ruled out by observing the absence of distal circulation and 40 ml 0.5% lidocaine is slowly injected through the intravenous cannula on the dorsum of the hand. The tourniquet remained inflated for 60 minutes from injection of lidocaine to reduce the risk of local anesthetic systemic toxicity (LAST)
  Other Names: Bier's Block
  Arms: Group A (Arm IVRA) 70 patients
Procedure: Forearm IVRA block — After placement of the forearm double tourniquet and exsanguination of the limb distal to the cuff by applying an Esmarch's bandage starting from the fingertips, the forearm tourniquet cuff is inflated to a pressure of 250 mmHg. The forearm tourniquet will be placed 5 cm distal to the medial epicondyle of the humerus and on the top of a circumferentially placed cotton cast. Subsequently, tourniquet failure is ruled out by observing the distal circulation and 25 ml 0.5% lidocaine is slowly injected through the intravenous cannula on the dorsum of the hand.
  Other Names: Mini Bier's Block
  Arms: Group F (Forearm IVRA) 70 patients

SUMMARY:
The technique of intravenous regional analgesia using a tourniquet consisting of two cuffs over the upper arm is a well-known procedure, With the tourniquet being conventionally placed over the upper arm, a relatively high dose of local anaesthetic drug is required and occasionally systemic toxic reactions have occurred.

The purpose of the present study is to establish the efficacy of the technique of intravenous regional analgesia with a forearm tourniquet using reduced doses of lidocaine.

DETAILED DESCRIPTION:
Several ways of anesthesia can be used to perform hand surgery, being general anesthesia, intravenous regional anesthesia as well as locoregional anesthesia. Locoregional anesthesia and intravenous regional anesthesia are often performed since patients can be discharged from the hospital more rapidly. A conventional Biers block is performed using a tourniquet on the upper arm to create a bloodless field and to contain the anesthetics within the surgical area.

A mini-Biers block in which the tourniquet is placed on the forearm, has been shown to be a safe and effective way of anesthesia to perform hand and wrist surgery. By using this type of anesthesia, the dose of the anesthetic can be reduced compared to a conventional Bier's block which reduces the risk of systemic toxicity reactions.

Intravenous regional anesthesia (IVRA) or Bier's Block is a simple and effective but underused anesthetic technique for hand and wrist surgery, This technique, introduced by Dr.August Bier in1908, provides complete anesthesia as well as a bloodless field during surgery.

Traditionally, an upper arm tourniquet has been used to sequester the local anesthetic and to create a bloodless Surgical field. Major complications after IVRA with an upper arm tourniquet are rare but are mostly related to local anesthetic systemic toxicity after release of the tourniquet.

Use of a forearm tourniquet has been introduced in 1978 and comes with the big advantage of lower (non-toxic) local anesthetic dosage requirement to produce a good quality of analgesia.

Consequently, there is no minimal tourniquet inflation time after forearm IVRA. In addition ,it has been postulated that sensory onset time after forearm IVRA may be shorter than after upper arm IVRA. With these two features forearm IVRA may be the ideal anesthetic technique for short surgery of hand and wrist.

ELIGIBILITY:
Inclusion Criteria:

* Patients of American Society of Anesthesiologists (ASA) physical status I to II.
* Both sexes.
* ≥ 21 to 65 years.
* scheduled for elective hand and wrist surgeries.

Exclusion Criteria:

* American society of Anesthesiologists (ASA) physical status ≥3 or BMI ≥40
* Patients will do bilateral hand surgery
* Local site infection.
* Allergy to local anesthetics.
* Patient refusal
* Patients with pre-existing myopathy or neuropathy on the operating limb.
* Patients with significant cognitive dysfunction.
* Chronic analgesic abuser patients.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
The primary aim of this study is to compare the analgesic effectivity of the arm intravenous regional anesthesia versus the forearm intravenous regional anesthesia. | surgery duration which is around 1.5 hour
  the analgesic effectivity of these techniques (graded as "complete" or "incomplete") and divide the effectivity in 4 grades. Grade 1 and grade 2 will be considered "complete" blockade, while grade 3 and grade 4 will be considered "incomplete" blockade. Grade 1: complete motor and sensory blockade. Grade 2: partial motor blockade but no pain. Grade 3: partial motor blockade with mild pain requiring rescue local or opioid analgesia. Grade 4: incomplete motor and sensory blockade requiring sedation/conversion to general anesthesia.

SECONDARY OUTCOMES:
Tourniquet time | From start of inflation until deflation of the tourniquet during surgery time which may last up to 90 minutes.
  Total time the tourniquet is inflated
Onset time of analgesia | At injection of the local anaesthetic until complete blockade of the sensory nerves during surgery
Tourniquet tolerance time | From start of inflation until deflation of the tourniquet during surgery
  Time required for the tourniquet to cause a painful sensation
Satisfaction with surgical conditions (bloodless field) | At the start of the surgical procedure
  Satisfaction with surgical conditions (bloodless field): assessed by the surgeon with a 5-point scale. This scale is ranged (1, 2, 3, 4, 5) in which 1 stands for "completely dissatisfied" and 5 for "completely satisfied".
Intraoperative pain score | Every 5 minutes up to 1.5 hours during the surgical procedure
  Intraoperative pain score
General satisfaction of the patient | Assessed on day 1 post surgery
  General satisfaction of the patient with the anesthesia technique (measured via a 7-point Likert scale, with 1 being completely dissatisfied and 7 being completely satisfied)
Postoperative pain score: Numeric Rating Scale(NRS) | Patients will be observed and data recording will be done every 2 hours for the first 24 hours for postoperative pain
  Postoperative pain score

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university hospitals, Cairo, Abbasia, Egypt